CLINICAL TRIAL: NCT00755755
Title: A Phase III, Randomized, Parallel Group, Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy and Safety of PGL4001 (Ulipristal) Versus Placebo for Pre-Operative Treatment of Symptomatic Uterine Myomas
Brief Title: PGL4001 Versus Placebo in Uterine Myomas
Acronym: PEARLI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGL07-021
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Uterine Myomas
MeSH Terms: interventions — ulipristal; Iron; ulipristal acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (PGL4001 5mg) (Experimental): PGL4001 5 mg (oral tablets) with concomitant oral administration of 1 tablet containing 80 mg Fe2+
  Interventions: Drug: PGL4001 (ulipristal) and iron
- B (PGL4001 10mg) (Experimental): PGL4001 10 mg (oral tablets) with concomitant oral administration of 1 tablet containing 80 mg Fe2+
  Interventions: Drug: PGL4001 (ulipristal) and iron
- C (placebo) (Placebo Comparator): PGL4001 matching placebo (oral tablets) with concomitant oral administration of 1 tablet containing 80 mg Fe2+
  Interventions: Drug: PGL4001 matching placebo and iron

INTERVENTIONS:
Drug: PGL4001 (ulipristal) and iron — tablets
  Other Names: Ulipristal acetate
  Arms: A (PGL4001 5mg)
Drug: PGL4001 matching placebo and iron — tablets
  Other Names: Placebo of ulipristal
  Arms: C (placebo)
Drug: PGL4001 (ulipristal) and iron — Tablets
  Other Names: Ulipristal acetate
  Arms: B (PGL4001 10mg)

SUMMARY:
This trial will assess the efficacy and safety of PGL4001 with concomitant iron administration versus placebo with concomitant iron administration, over a 3-month period for the pre-operative treatment of pre-menopausal women suffering from excessive uterine bleeding due to uterine myoma.

ELIGIBILITY:
Inclusion Criteria:

* Be a pre-menopausal woman between 18 and 50 years inclusive.
* Have excessive uterine bleeding due to myoma.
* Have a myoma-related anaemia.
* Have a myomatous uterus with at least one myoma of ≥ 3 cm diameter in size.
* Be eligible for one surgical procedure: e.g. hysterectomy, myomectomy or others.
* If of childbearing potential the subject must be practicing a non-hormonal method of contraception.
* Have a Body Mass Index (BMI) ≥ 18 and ≤ 40.

Exclusion Criteria:

* Has a history of or current uterine, cervical, ovarian or breast cancer.
* Has a history of or current endometrium atypical hyperplasia.
* Has a known severe coagulation disorder.
* Has a history of or current treatment for myoma with a Selective Progesterone Receptor Modulator (SPRM) or a GnRH-agonist.
* Has abnormal hepatic function at study entry.
* Has a positive pregnancy test at baseline or is nursing or planning a pregnancy during the course of the study.
* Has a current (within twelve months) problem with alcohol or drug abuse.
* Is currently enrolled in an investigational drug or device study or has participated in such a study within the last 30 days.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 241 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Elke Bestel, Study Director — PregLem SA
Locations (38):
- Czechia (4):
  - Gynekologicko-porodnicka klinika FN Brno, Brno
  - Mediva, Prague
  - Gynekologicko-porodnicka klinika 1.LF UK a VFN, Prague
  - Gynekologicko-porodnicka klinika UK 2.LF a FN, Prague
- Hungary (6):
  - Rethy-Pal Hospital-Clinic Bekescsaba, Department of Obstetrics and Gynecology, Békéscsaba
  - Saint Stephen Hospital of Budapest,Department of Obstetrics, Gynecology and Gynecological Oncology, Budapest
  - Fovarosi Bajcsy-Zsilinszky Hospital, Department of Obstetrics and Gynecology, Budapest
  - Dr. Bugyi Istvan Hospital, Department of Obstetrics and Gynecology, Szentes
  - Saint George Hospital of Fejer County, Department of Obstetrics and Gynecology, Székesfehérvár
  - Saint Borbala Hospital of Komarom-Esztergom County, Department of Obstetrics and Gynecology, Tatabánya
- India (6):
  - Dr. Jilla Hospital, Aurangabad
  - M. S. Ramaiah Medical College and Memorial Hospital, Bangalore
  - Divakars Speciality Hospital, Bangalore
  - Sri Ramachandra Medical College and Research Institute, Chennai
  - Om Women's Hospital, Nagpur
  - Nagpur Test Tube Baby Centre, Nagpur
- Romania (6):
  - Central Medical Sanador, Bucharest
  - Departamentul de Obstretica Ginecologie si Nou Nascuti, Bucharest
  - Centrul Medical Euromed, departementul de Obstetrica/Ginecologie, Bucharest
  - Sectia Obstretica-Ginecologie Spitalul Clinic Dr. Ioan Cantacuzino, Bucharest
  - Spitalul Clinic de Obstetrica Ginecologie Oradea, Oradea
  - Spitalul Clinic Judetean de urgenta, sectia de obstetrica Ginecologie I, Târgu Mureş
- Russia (9):
  - Northern State Medical University, Arkhangelsk
  - Kursk State Medical University, Kursk
  - American Medical Clinic, Saint Petersburg
  - Saint-Petersburg City Alexandrovsky Hospital, Saint Petersburg
  - Military Medical Academy n.a.S.M Kirov, chair of Obstetrics and Gynecology, Saint Petersburg
  - Medical Research Institute (MRI), Saint Petersburg
  - Russian Scientific Research Center of Radiology and Surgical Technologies, Saint Petersburg
  - Scientific Research Institute of Obstetrics and Gynecology n.a. D.O.Ott of RAMS, Saint Petersburg
  - OAO "Medical company IDK", Samara
- Ukraine (7):
  - Donetsk National Medical University, Department of Obstetrics, Gynecology and Perinatology FPE, Donetsk
  - City Clinical Hospital N9, Kiev
  - Institute of Pediatrics, Obstetrics and Gynecology, Department of Endocrine Gynecology, Kiev
  - Kiev Maternity Hospital No.2, Kiev
  - State Enterprise "Institute of Pediatrics, Obstetrics and Gynecology of AMS of Ukraine, Kyiv
  - Lviv National Medical University named after Danylo Halytskyy, Lviv
  - Medical Sanitory Centre VAT "Motor Sich" Gynecology department, Zaporizhzhya

REFERENCES:
- [Result] Donnez J, Tatarchuk TF, Bouchard P, Puscasiu L, Zakharenko NF, Ivanova T, Ugocsai G, Mara M, Jilla MP, Bestel E, Terrill P, Osterloh I, Loumaye E; PEARL I Study Group. Ulipristal acetate versus placebo for fibroid treatment before surgery. N Engl J Med. 2012 Feb 2;366(5):409-20. doi: 10.1056/NEJMoa1103182. PMID 22296075
- [Derived] Barlow DH, Lumsden MA, Fauser BC, Terrill P, Bestel E. Individualized vaginal bleeding experience of women with uterine fibroids in the PEARL I randomized controlled trial comparing the effects of ulipristal acetate or placebo. Hum Reprod. 2014 Mar;29(3):480-9. doi: 10.1093/humrep/det467. Epub 2014 Jan 23. PMID 24457604

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (Placebo)
Started | 95 (Safety population) | 98 (Safety population) | 48 (Safety population)
Completed | 89 (Patients who completed the overall study up to the follow-up visit (visit 6)) | 90 (Patients who completed the overall study up to the follow-up visit (visit 6)) | 45 (Patients who completed the overall study up to the follow-up visit (visit 6))
Not Completed | 6 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (Placebo) | Total
Number analyzed (Participants) | 95 | 98 | 48 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 95 | 98 | 48 | 241
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.2 (5.9) | 42.0 (5.5) | 41.6 (5.6) | 41.6 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 98 | 48 | 241
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czech Republic | 7 | 6 | 3 | 16
  Hungary | 7 | 11 | 9 | 27
  India | 10 | 11 | 7 | 28
  Romania | 17 | 17 | 8 | 42
  Russian Federation | 28 | 19 | 13 | 60
  Ukraine | 26 | 34 | 8 | 68

OUTCOME MEASURES:

1. Primary Outcome: Co-primary Endpoint: Percentage of Subjects With Reduction in Uterine Bleeding Defined as a Pictorial Blood-loss Assessment Chart (PBAC) Score <75 at End-of-treatment Visit (Week 13)
Description: Uterine bleeding was assessed with the use of the PBAC, a validated self-reporting method to estimate menstrual blood loss.
  Patients recorded daily the number of tampons and towels used and the degree to which individual items were soiled with blood (plus small or large clots). Monthly scores range from 0 (amenorrhea) to more than 500, with higher numbers indicating more bleeding.
  A slightly stained tampon/towel scores 1, a partially stained tampon/towel scores 5, a completely saturated tampon scores 10 and a completely saturated towel scores 20. Small clots/flooding (2cm) score 1. Large clots/flooding (3cm) score 5.
  Menorrhagia is defined as a PBAC > 100 during one menstrual period which approximates to a blood loss of > 80 mL. A PBAC of 400 corresponds to a blood loss of around 300 mL or approximately 80 tampons/towels used.
  The week 13 PBAC score was calculated using the last 28 days of treatment.
Time Frame: Week 13 visit
Population: Intent-to-treat
Measure: Number; unit: percentage of patients
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (Placebo)
Number analyzed (Participants) | 94 | 93 | 48
percentage of patients | 91.5 | 92.5 | 18.8
Statistical Analysis 1: Comparison: A (PGL4001 5mg) vs C (Placebo); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — As comparison involved two doses of PGL4001 vs Placebo, Bonferroni correction used with p-values doubled (threshold was 0.05) and confidence intervals adjusted; Adjustment for randomization strata; Difference in proportions = 72.7, 95% CI 2-sided [55.1 to 83.2] — Confidence intervals with the use of Newcombe-Wilson score method (uncorrected)
Statistical Analysis 2: Comparison: B (PGL4001 10mg) vs C (Placebo); Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — As comparison involved two doses of PGL4001 vs Placebo, Bonferroni correction used with p values doubled (threshold was 0.05) and confidence intervals adjusted; Adjustment for randomization strata; Difference in proportions = 73.7, 95% CI 2-sided [56.2 to 84.0] — Confidence intervals with the use of Newcombe-Wilson score method (uncorrected)

2. Primary Outcome: Co-primary Endpoint: Percent Change in Total Myoma Volume Assessed by Magnetic Resonance Imaging (MRI) From Screening to End of Treatment Visit (Week 13 Visit)
Description: Percent change in total fibroid volume from screening to end of treatment visit (Week 13 visit) assessed by MRI and read centrally by a radiologist who was unaware of the study-group assignments. The total fibroid volume was the sum of the individual fibroid volumes.
Time Frame: Week 13
Population: Intent-to-treat
Measure: Median (Full Range); unit: percentage of change
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (Placebo)
Number analyzed (Participants) | 85 | 80 | 45
percentage of change | -21.2 [-100 to 223.4] | -12.3 [-100 to 146.6] | 3 [-100 to 134.8]
Statistical Analysis 1: Comparison: A (PGL4001 5mg) vs C (Placebo); Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 1]; Use of the Van Elteren extension to the Wilcoxon rank-sum test with adjustment for randomization strata; Median Difference (Final Values) = -22.6, 95% CI 2-sided [-36.1 to -8.2] — Hodges-Lehmann point estimator with corresponding Moses confidence interval
Statistical Analysis 2: Comparison: B (PGL4001 10mg) vs C (Placebo); Test type: Superiority or Other; p = 0.006, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 1, analysis 2]; Use of the Van Elteren extension to the Wilcoxon rank-sum test with adjustment for randomization strata; Median Difference (Final Values) = -18.2, 95% CI 2-sided [-33.0 to -5.2] — Hodges-Lehmann point estimator with corresponding Moses confidence interval

ADVERSE EVENTS:
Time Frame: 3 years 2 months
Arm/Group | A (PGL4001 5mg) | B (PGL4001 10mg) | C (Placebo)
Serious Adverse Events (participants affected / at risk) | 2/95 | 1/98 | 2/48
Other Adverse Events (participants affected / at risk) | 47/95 | 52/98 | 22/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (PGL4001 5mg) (N=95) | B (PGL4001 10mg) (N=98) | C (Placebo) (N=48)
Ovarian hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
New uterine leiomyoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
breast cancer (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A (PGL4001 5mg) (N=95) | B (PGL4001 10mg) (N=98) | C (Placebo) (N=48)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 3 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 4 (6) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (6) | 10 (19) | 2 (2)
Breat pain / tenderness / disconfort (Reproductive system and breast disorders) | 2 (2) | 6 (6) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 4 (4) | 0 (0)
Hypercholesterolemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (2) | 2 (2)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 14 (18) | 14 (16) | 6 (10)
Nervous system disorders (Nervous system disorders) | 4 (7) | 11 (22) | 3 (4)
Infections and infestations (Infections and infestations) | 8 (8) | 12 (15) | 3 (4)
Endocrine disorders (Endocrine disorders) | 5 (8) | 8 (8) | 1 (2)
General disorders and administration site conditions (General disorders) | 5 (5) | 4 (4) | 2 (3)
Diziness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 7 (10) | 4 (4) | 2 (3)
Gastrointestinal disorders (Gastrointestinal disorders) | 9 (16) | 10 (13) | 3 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No